CLINICAL TRIAL: NCT01217853
Title: Comparison of 24-hour Continuous IOP Monitoring With a Contact Lens-based Sensor to Goldmann Applanation Tonometry
Brief Title: 24h Continuous Intraocular Pressure (IOP) Monitoring vs Goldmann Applanation Tonometry
Status: Completed | Type: Observational
Sponsor: Sensimed AG (Industry)
Collaborators: Schlossparkklinik (Unknown)
Responsible Party: Jean-Marc Wismer, Sensimed AG
Other Study IDs: 09/10
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SENSIMED Triggerfish
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish — Contact lens-based device for continuous intraocular pressure monitoring

SUMMARY:
A study in which intraocular pressure (IOP) will be monitored over 24 hours using the SENSIMED Triggerfish® device and Goldmann applanation tonometry (GAT) in primary open angle glaucoma patients. The aim of this study is to investigate the comparability of diurnal IOP patterns emerging from SENSIMED Triggerfish and GAT.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for the investigation
* Patients with primary open angle glaucoma (POAG), defined as open angle ≥ 30°, confirmed visual field loss (Mean Defect/Least Variance ≤ 2dB) and/or optic nerve head damage (cup disc ratio > 0,5)
* Age 40-70 years at inclusion
* Not more than 4 diopters spherical equivalent on the study eye
* Not more than 2 diopters cylinder equivalent on the study eye
* For women of childbearing potential, adequate contraception
* Stable anti-glaucomatous therapy 4 weeks before the first 24-hour IOP assessment session and throughout the investigation

Exclusion Criteria:

* Patients not able to understand the character and individual consequences of the investigation
* Patients committed to an institution by virtue of an order issued either by the courts or by an authority
* Absence of or withdrawn informed consent
* Patients with contraindications for silicone contact lens wear
* Wear of full frame metallic glasses during SENSIMED Triggerfish monitoring
* Eye disorders including severe dry eye
* Eye disorders secondary to POAG
* Patient who have had ocular surgery within the last 3 months
* Corneal or conjunctival abnormality or irregularity hindering correct contact lens adaptation
* Pregnancy and lactation
* Allergy to oxybuprocaine (ocular anesthesia)
* Simultaneous participation in other clinical research

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients 40 to 70 years old and diagnosed with primary open angle glaucoma.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
SENSIMED Triggerfish output values | During 24 hours
  Patients will undergo one session of 24-hour SENSIMED Triggerfish continuous intraocular pressure monitoring in one eye.
Goldmann applanation tonometry values | During 24 hours
  Goldmann applanation IOP readings will be done in the other eye at regular intervals during 24-hour SENSIMED Triggerfish IOP monitoring and in both eyes during another 24-hour session.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Erb, Prof, Principal Investigator — Schlosspark-Klinik Berlin
Locations (2):
- Germany (2):
  - Schlosspark-Klinik, Berlin
  - Johannes Gutenberg Universitätsklinik Mainz, Mainz